CLINICAL TRIAL: NCT02108249
Title: Annex™ Adjacent Level System for Treatment of Adjacent Level Disease
Status: Completed | Type: Observational
Sponsor: Spine Wave (Industry)
Responsible Party: Sponsor
Other Study IDs: SW-ANX1401
Record Dates: First submitted 2014-04-02; First posted 2014-04-09 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Degenerative Disc Disease; Adjacent Level Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Annex Group: Patients prospectively treated with Annex™ Adjacent Level System
  Interventions: Device: Annex™ Adjacent Level System
- Retrospective Control: Patients previously treated for adjacent level disease using other systems

INTERVENTIONS:
Device: Annex™ Adjacent Level System
  Groups: Annex Group

SUMMARY:
The purpose of this study is to evaluate the clinical, radiological, and surgical outcomes of the Annex™ Adjacent Level System for the treatment of adjacent level disease of the lumbar spine. The Annex™ Adjacent Level System is a spinal fixation system intended to be used with commercially available pedicle screw fixation systems in order to extend existing pedicle screw constructs. Subjects will be evaluated over a 2 year period and compared to historical control.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18-85 years of age
* Single level adjacent level segment disease (ALD) in the lumbar spine (L1-S1).

Exclusion Criteria:

* trauma, tumor, pseudoarthrosis, revision, or same-level recurrent stenosis
* cervical fusion candidates
* extraspinal cause of back pain
* local or systemic infection
* pregnant / able to become pregnant and not following a reliable contraceptive method
* Severe osteoporosis or osteopenia
* Morbid obesity defined as BMI > 40
* Anatomy or other factors that prohibit safe surgical access to the surgical site
* Allergy or sensitivity to any component of the treatment procedure
* Inadequate tissue coverage over the operative site
* Inadequate bone stock or bone quality
* Fever or leukocytosis
* Uncorrectable coagulopathy or hemorrhagic diathesis
* Cardiopulmonary conditions that present prohibitive anesthesia risk
* Neuromuscular disease or disorder
* Mental illness
* Has an active workman's compensation claim

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population for both the treatment and control groups will include adult (skeletally mature) men and women who were previously implanted with rigid posterior fixation (pedicle screw/rod constructs) in the thoracolumbar spine and who later developed adjacent level disease (ALD) at a lumbar level.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
% Improvement in Operative/Discharge parameters including surgical time and hospital stay | within 30 days after treatment
Surgical Complication rate compared to retrospective chart review | Within 30 days of treatment

SECONDARY OUTCOMES:
% Pain reduction on VAS | Up to 2 years post-treatment
% Improvement in Disability using ODI | Up to 2 years post-treatment
% Improvement in Quality of Life using SF-36 | Up to 2 years post-treatment
% Patient Satisfaction with procedure | Up to 2 years post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Carolinas Neurosurgery and Spine, Charlotte, North Carolina, United States